CLINICAL TRIAL: NCT05811221
Title: Application of Different Modes of Esketamine Administration in Pediatric Day Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Wang wanxia, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-YKL01-（ke11）
Record Dates: First submitted 2023-03-01; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Pain
Keywords: Pediatric circumcision; Mode of administration; Day surgery; Esketamine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single group (Active Comparator): give esketamine 0.75 mg/kg at the time of induction
  Interventions: Drug: Esketamine of single injection
- intermittent group (Experimental): give esketamine 0.5mg/kg during anesthesia induction, and during the measuring ring esketamine 0.25mg/kg was given again
  Interventions: Drug: Esketamine of Intermittent injection

INTERVENTIONS:
Drug: Esketamine of single injection — Single group: give esketamine 0.75 mg/kg at the time of induction
  Other Names: A single injection of esketamine at the time of anesthesia induction
  Arms: single group
Drug: Esketamine of Intermittent injection — Intermittent group: give esketamine 0.5mg/kg during anesthesia induction, and during the measuring ring esketamine 0.25mg/kg was given again
  Other Names: A Intermittent injection of esketamine at the time of anesthesia induction
  Arms: intermittent group

SUMMARY:
To explore the application of different administration modes of esketamine in pediatric day circumcision, in order to find an anesthesia scheme more suitable for day pediatric circumcision.

DETAILED DESCRIPTION:
The current clinical study believes that esketamine is suitable for pediatric anesthesia because of its advantages of light respiratory depression, low secretions, low incidence of psychomotor reactions and fast recovery of anesthesia, but there are few related studies on its administration mode and timing in clinical application, this study aims to explore the application of different administration methods of esketamine in pediatric day circumcision, and find an anesthesia scheme more suitable for day circumcision, in order to provide new ideas for anesthesia for pediatric day circumcision.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I and II children
* Age 5-12 years
* Foreskin cerclage is proposed
* No history of upper respiratory tract infection in the past two weeks
* Obtain the consent of the child's family

Exclusion Criteria:

* Hepatic and renal insufficiency, coagulation dysfunction
* Those who are allergic to esketamine
* History of cognitive impairment
* epilepsy
* other psychiatric and neurological disorders

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-04-02 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
One-time success rate of anesthesia | During surgery
  No movement during anesthesia

SECONDARY OUTCOMES:
Systolic blood pressure | During surgery
  Systolic blood pressure
Diastolic blood pressure | During surgery
  Diastolic blood pressure
Heart rate | During surgery
  Heart rate
intraoperative propofol dosage, esketamine dosage | During surgery
  intraoperative propofol dosage, esketamine dosage
Duration of surgery | During surgery
  Duration of surgery
Time to open eyes | During surgery
  Time to open eyes
Time to talk | During surgery
  Time to talk
VAS(visual analogue scale) score | 12 hours after the end of surgery
  A score to assess pain, use a swimming ruler about 10 cm long, marked with 10 scales on one side, with "0" and "10" ends at each end, 0 points means no pain, and 10 points represent the most severe pain that is unbearable.
Incidence of adverse effects (hypotension, hypertension, respiratory depression, postoperative pain, diplopia, mania) | 12 hours after the end of surgery
  Incidence of adverse effects (hypotension, hypertension, respiratory depression, postoperative pain, diplopia, mania)